CLINICAL TRIAL: NCT07241455
Title: Validity of the Children's Chelsea Critical Care Physical Assessment Tool (cCPAx-TR) in Turkish Pediatric Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ayse Asik, Pediatric Critical Care Fellow, Department of Pediatrics, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: cCPAxTR2025V1
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Critical Illness; Physical Function Assessment; Functional Status; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center, prospective observational study aims to translate, culturally adapt, and evaluate the validity and reliability of the Children's Chelsea Critical Care Physical Assessment Tool (cCPAx) in Turkish pediatric intensive care settings (cCPAx-TR). We will assess content validity with an expert panel, feasibility in a pilot run, test-retest reliability, internal consistency, and criterion validity against established clinical scores.

DETAILED DESCRIPTION:
This single-center, prospective observational study aims to translate, culturally adapt, and evaluate the Turkish version of the Children's Chelsea Critical Care Physical Assessment Tool (cCPAx-TR) for use in pediatric intensive care settings.

The study will be conducted in the Pediatric Intensive Care Unit (PICU) of Göztepe Prof. Dr. Süleyman Yalçın City Hospital. The translation and cultural adaptation will follow internationally accepted guidelines, including forward and backward translation, expert panel review, and pilot testing.

Following pilot testing, psychometric evaluation will include assessments of internal consistency, test-retest reliability, and criterion validity by comparison with established clinical scores such as the Functional Status Scale (FSS), Glasgow Coma Scale (GCS), and Pediatric Logistic Organ Dysfunction (PELOD) score. Feasibility and safety will be analyzed based on completion rate, administration time, and occurrence of adverse events.

The study population will include children aged 2-18 years who are admitted to the PICU and are clinically stable enough for bedside physical function assessment.

ELIGIBILITY:
Inclusion Criteria

* Children aged 2 to 18 years
* Admitted to the pediatric intensive care unit (PICU)
* Clinically stable for bedside assessment
* Parental or guardian informed consent obtained (and child assent when appropriate)
* Able to perform or be observed for at least one item of the cCPAx-TR
* Exclusion Criteria
* Unstable hemodynamics or severe hypoxemia that prevents safe assessment
* Deep sedation or neuromuscular blockade that prevents observation at both assessments
* Severe orthopedic or neurological conditions (for example, unstable fractures or acute paralysis) that prohibit safe mobilization
* Expected death or withdrawal of care within 24 hours
* Refusal of consent by parents or guardians

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include pediatric patients aged 2 to 18 years who are admitted to the pediatric intensive care unit (PICU) at Göztepe Prof. Dr. Süleyman Yalçın City Hospital. The study population represents critically ill children with various underlying medical, surgical, and neurological conditions who are clinically stable enough to undergo bedside physical function assessment. Both intubated and non-intubated patients will be eligible for inclusion, provided that they meet stability and safety criteria for evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Test-retest intraclass correlation coefficient (ICC) - total cCPAx-TR score | two measurements conducted 48 hours apart
  The intraclass correlation coefficient (two-way mixed, absolute agreement) for the cCPAx-TR total score between two assessments administered 48 hours apart in clinically stable participants.

CONTACTS AND LOCATIONS:
Overall Officials: Muhterem Duyu, Study Chair
Locations (1):
- Göztepe Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Kadıkoy, Turkey (Türkiye)